CLINICAL TRIAL: NCT05065632
Title: Population-based Age-stratified Seroepidemiological Investigation of Coronavirus 2019 (COVID-19) Infection in Gabon
Brief Title: Seroepidemiological Investigation of Coronavirus 2019 (COVID-19) Infection in Gabon
Acronym: Sero-CoV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prof. Ayola Akim ADEGNIKA (Other)
Responsible Party: Sponsor-Investigator, Prof. Ayola Akim ADEGNIKA, Prof. Dr, Centre de Recherche Médicale de Lambaréné
Organization: Centre de Recherche Médicale de Lambaréné (Other)
Other Study IDs: 0056/2021/P/SG/CNER
Record Dates: First submitted 2021-09-30; First posted 2021-10-04 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Laboratory Confirmed SARS-CoV-2 Infection Without Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Venous Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Groupe 1: [1-15[
  Interventions: Diagnostic Test: Wantai kit Elisa
- Group 2: [15- 30[
  Interventions: Diagnostic Test: Wantai kit Elisa
- Group 3: [30-45[
  Interventions: Diagnostic Test: Wantai kit Elisa
- Group 4: [45-60[
  Interventions: Diagnostic Test: Wantai kit Elisa
- Group 5: 60+
  Interventions: Diagnostic Test: Wantai kit Elisa

INTERVENTIONS:
Diagnostic Test: Wantai kit Elisa — to mesure antibodies against SARSCov-2 recombinant antigen

SUMMARY:
Gabon is the 3rd country most affected by COVID-19 behind Cameroon and Democratic Republic of Congo in Central Africa, with 8860 cases and 54 deaths in critically ill patients, since the first confirmed case of COVID-19 on the 10th of March 2020 (https://africacdc.org/covid-19/). Most of the individuals infected by SARS-CoV-2 are asymptomatic and they represent a major source of viral spread. To date, African countries have been less affected by deaths caused by the Covid-19 pandemic compared to other countries. It is currently unknown why Africa has avoided more deaths and appears to not simply be due to a lack of testing, since the overall death rate has not increased. Better quality data on seroprevalence in different African regions and proven explanations of the differences between Africa and other continents, are urgently needed. The aim of this study is to learn about the proportion of people after a first pic of transmission, who have been exposed to COVID-19 in Gabon by testing for plasma antibodies to the SARS-CoV-2 virus.

The overall goal of this study is to examine the trend of specific anti-SARS-CoV-2 antibodies in Gabonese population.

DETAILED DESCRIPTION:
Based on its technical capacities (ELISA bench and multiparametric flow cytometer), we will provide evident data on the immune responses in Covid-19 infected patients. The quantification of antibodies against SARS-CoV-2 recombinant protein will be done by ELISA using Wantai ELISA total Ab. Meanwhile, data on clinical status will be recorded and classified using WHO patient form. Data obtained will be analyzed by a statistician based at CERMEL using robust models in compliance with the type of data generated.

ELIGIBILITY:
Inclusion Criteria:

* Persons of both sexes aged one year and older and residing for more than three months in the study area are eligible to participate in the study

Exclusion Criteria:

* Any person not residing in the locality surveyed or any person residing for less than three months. Refusal to give informed consent and contraindication to venipuncture venipuncture.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 3455 people living in Gabon, aged from 1 year, and above will be stratified by age and included in this study
Sampling Method: Probability Sample
Enrollment: 3455 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
seroprevelence on SARS-Cov- 2 infection in Gabon | 4 Months
  assess the specific anti-SARS-CoV-2 antibodies in individuals and for modeling the evolution of the COVID-19 outbreak.

CONTACTS AND LOCATIONS:
Overall Officials: Ayola Akim A ADEGNIKA, PhD, Principal Investigator — Centre de Recherche Médicale de Lambaréné
Locations (1):
- Centre de Recherches Medicales de Lambarene, Lambaréné, Gabon

IPD SHARING:
Plan to Share IPD: No